# **Statistical Analysis Plan**

## **Official Title**:

Effectiveness of a Multimodal Information Technology-enhanced Hand Hygiene Improvement Strategy on Healthcare-associated Infections in Nursing Homes

**NCT Number**:

NCT06925620

**Document Date:** 

January 27, 2022

#### **Statistical Analysis Plan**

### **Study Title**:

Effectiveness of a Multimodal Information Technology-enhanced Hand Hygiene Improvement Strategy on Healthcare-associated Infections in Nursing Homes

### **Objectives**:

- 1. To determine whether the multimodal hand hygiene program improves knowledge, compliance, and technique accuracy.
- 2. To evaluate the reduction in HAI density following the intervention.

Analysis Population: All participants enrolled and completing baseline assessments.

#### **Statistical Methods:**

- 1. **Descriptive Statistics**: Means, standard deviations, frequencies, and percentages for baseline characteristics.
- 2. Comparative Analysis:
  - (1) Generalized Estimating Equations (GEE) to compare compliance, accuracy, and knowledge scores over time between groups.
  - (2) Incidence density of HAI compared using rate ratios.
- 3. **Significance Level**: Two-tailed p-value < 0.05 will be considered statistically significant.

**Handling of Missing Data**: Missing data will be addressed using multiple imputation if applicable.

**Software**: IBM SPSS Statistics Version 26.0.